CLINICAL TRIAL: NCT06246409
Title: Modernizing Instructions to Improve Treatment Participation of Subjects During Their First Radiotherapy
Acronym: PEERs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UF-CCPS-038; IRB202401379 (Other: University of Florida)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: patient comfort; patient participation; external beam radiotherapy; radiation oncology
MeSH Terms: conditions — Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Existing patient instructions (Active Comparator)
  Interventions: Behavioral: Existing patient instructions
- Arm 2: Modernized patient instructions (Experimental)
  Interventions: Behavioral: Modernized patient instructions

INTERVENTIONS:
Behavioral: Modernized patient instructions — Patients will be given modernized patient instructions prior to radiotherapy treatment.
  Arms: Arm 2: Modernized patient instructions
Behavioral: Existing patient instructions — Patients will be given the patient instructions currently in use prior to radiotherapy treatment.
  Arms: Arm 1: Existing patient instructions

SUMMARY:
Daily patient participation is critical to the successful, life-saving delivery of radiotherapy. There is very little in the literature describing the best way to prepare patients to give optimal participation. This study aims to look at an already-prepared conversion of patient instruction materials and measure whether the improvement in clarity and specificity produces the desired changes in patient decision-making and emotional comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old planning their first external beam radiotherapy
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.

Exclusion Criteria:

* Have received external beam radiotherapy in the past
* External beam radiotherapy is initiated as inpatient.
* External beam radiotherapy consists of less than 3 fractions.
* Planned radiotherapy that does not employ an external beam
* Planned participation in a clinical study that prohibits participation in a second, concurrent treatment trial
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Unintentional missed treatment days | 8 weeks
  Determine the number of unintentional missed days of treatment during a course of radiotherapy

SECONDARY OUTCOMES:
Patient-reported comfort | 8 weeks
  Evaluate patient-reported comfort with participation in radiotherapy.
Unplanned clinic visits | 8 weeks
  Determine the average number of unplanned clinic visits during radiotherapy.
Emergency department visits | 8 weeks
  Determine the average number of emergency department visits during radiotherapy.
Hospitalizations | 8 weeks
  Determine the average number of hospitalizations during radiotherapy.
Rate of treatment completion | 8 weeks
  Determine the rate of completion of the prescribed number of radiotherapy treatments.
Patient participation in treatment | 8 weeks
  Determine the percentage of patients fully participating in their radiotherapy treatment, as assessed by Likert scale ratings given by the therapist. Patients will be rated by the therapist on factors such as correct patient-initiated alignment of body, holding still, and following breath-hold directions.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Hitchcock, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States